CLINICAL TRIAL: NCT03186274
Title: Discussing Death and Dying: An End of Life Curriculum to Empower Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Katherine Schultz, Resident, Department of Pediatrics, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 170675
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Education, Medical; Education, Medical, Graduate; Care, Palliative; Medicine, Palliative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Those in the control group (CG) will write a pre and post-study reflection essay discussing their experiences with end of life discussions.
- Facilitated Group Session (Experimental): Participants in Facilitated Group Session (previously called Intervention Group 1) will watch a pre-recorded video describing the SPIKES model and then take part of a facilitated guided group session reviewing the model and group interview of standardized/simulated patient encounter.
  Interventions: Behavioral: Facilitated Group Session
- CELA Session (Experimental): Participants in the CELA Session (previously called Intervention Group 2) will watch a pre-recorded video describing the SPIKES model and then participate in an individualized standardized/simulated patient scenario that will be filmed at the Center for Experiential Learning and Assessment (CELA).
  Interventions: Behavioral: CELA Session

INTERVENTIONS:
Behavioral: Facilitated Group Session — Participants will review the SPIKES model with a facilitator and then participate in a guided and supported simulated patient encounter utilizing aspects of the SPIKES model, with feedback at the end of the session.
  Arms: Facilitated Group Session
Behavioral: CELA Session — Participants will review the SPIKES model on their own and then participate in a simulated patient encounter utilizing the SPIKES model. They will receive feedback following the encounter.
  Arms: CELA Session

SUMMARY:
This study will evaluate how the educational intervention utilized affects pediatric resident comfort level with EOL discussions.

DETAILED DESCRIPTION:
One of the most challenging roles a physician can serve is delivering life altering and/or bad news to patients and their families, and yet this skill is not widely taught to physicians. A survey from 2003 of pediatric residents found that not only was there minimal education and training in this area, but that they felt there was no natural improvement in their skills from the first to third year of training. It has also been shown that the art of eliciting a patient or family's concerns about death and responding to them is felt to be poorly taught. Worse, residents have indicated that a hidden curriculum in medicine seems to indicate that there is no value to these conversations at all. Residents are not the only stakeholders involved who have expressed concern with this reality. Parents of pediatric patients have repeatedly reported wanting increased sensitivity and clarity during sharing of life-altering information. Up to 75% of parents have reported a negative experience involving end of life (EOL) discussions, and cited inexperience, lack of comfort in communication, and a lack of knowledge as contributing factors to their negative experiences. Less than 18% of students and residents report receiving formal education in EOL discussions, despite the fact that 90% or more of residents have identified caring for those dying as part of a physician's responsibilities. Of residents who do get experience with EOL discussions, less than 2/3 receive feedback. Some residencies, such as internal medicine, have recognized the need for formal instruction on how to have EOL discussions is needed and have implemented formal programs to answer it, and it has even become a standard expectation for many fellowships. Formal education regarding EOL has also become a standard expectation for many fellowships, including pediatric neonatology, intensive care, and hematology/oncology. Despite the evidence that there is need for formal intervention and education regarding EOL care, there has been little advancement towards implementing a formal curriculum in pediatric residency programs. Review of the literature demonstrates that only one study has developed a formal curriculum involving a method called SPIKES (Setting, Perception, Involvement, Knowledge, Empathy, and Summary) that targets pediatric residents. The initial data from this study is promising and indicates increased comfort level in residents. However, to date no study has evaluated if the method of instruction affects the resident education, an important consideration as some interventions (ex. standardized patients) are more costly and time consuming than others (ex. facilitator guided small group sessions).

ELIGIBILITY:
Inclusion Criteria:

* Post Graduate Year (PGY) 2 or PGY-3 resident participating in the already-required Advocacy rotation at Monroe Carrell Jr. Children's Hospital at Vanderbilt
* Availability to participate in self reflection essays and simulated patient case
* English speaking

Exclusion Criteria:

* Medical students, PGY-1, PGY-4 or PGY-5 residents, fellows or learners not participating in the already-required Advocacy rotation
* Inability to participate in self reflection essays and simulated patient case
* Non-English speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Self-reported resident competency | 1 year
  Residents will complete validated pre- and post-surveys to evaluate their competency in having end of life discussions. The scale is 1-4, where 1 indicates very comfortable and 4 indicates very uncomfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Travis Crook, MD, Study Chair — Pediatric Hospital Medicine
Locations (1):
- Monroe Carell Junior Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tait GR, Hodges BD. Residents learning from a narrative experience with dying patients: a qualitative study. Adv Health Sci Educ Theory Pract. 2013 Oct;18(4):727-43. doi: 10.1007/s10459-012-9411-y. Epub 2012 Oct 6. PMID 23053870
- [Background] Wolfe AD, Denniston SF, Baker J, Catrine K, Hoover-Regan M. Bad News Deserves Better Communication: A Customizable Curriculum for Teaching Learners to Share Life-Altering Information in Pediatrics. MedEdPORTAL. 2016 Aug 12;12:10438. doi: 10.15766/mep_2374-8265.10438. PMID 31139729
- [Background] Sullivan AM, Lakoma MD, Block SD. The status of medical education in end-of-life care: a national report. J Gen Intern Med. 2003 Sep;18(9):685-95. doi: 10.1046/j.1525-1497.2003.21215.x. PMID 12950476
- [Background] Keefer P, Pituch K, Murphy T, et al. A child's last hours - multidisciplinary training in end-of-life care for professionals working in children's hospitals: newborn with lethal congenital anomalies. MedEdPORTAL Publications. 2015;11:10108. http://doi.org/10.15766/mep_2374-8265.10108
- [Background] Rock L, Gadmer N, Arnold R, et al. Critical care communication skills training for internal medicine residents. MedEdPORTAL Publications. 2015;11:10212. http://doi.org/10.15766/mep_2374-8265.10212
- [Background] Brock K, Cohen H, Sourkes B, et al. Teaching pediatric fellows palliative care through simulation and video intervention: a practical guide to implementation. MedEdPORTAL Publications. 2015;11:10284. http://doi.org/10.15766/mep_2374-8265.10284
- [Background] Brown C, Gephardt G, Lloyd C, Swearingen C, Boateng B. Teaching palliative care skills using simulated family encounters. MedEdPORTAL Publications. 2011;7:8507. http://doi.org/10.15766/mep_2374-8265.8507
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Jackson J, Albertini L. Caring for children with chronic health care needs: an introductory curriculum for pediatric residents. MedEdPORTAL Publications. 2012;8:9172. http://doi.org/10.15766/mep_2374-8265.9172
- [Background] Mintzer M, Chen A, Conway Copper T, et al. Breaking bad news using role playing: a multimedia instructional activity for teaching medical trainees. MedEdPORTAL Publications. 2014;10:9798. http://doi.org/10.15766/mep_2374-8265.9798
- [Background] Reichert J, Parmelee D, Bognar S, Durgans K, Godoy M. A LION IN THE HOUSE module for health care education: pediatric end-of-life case studies. MedEdPORTAL Publications. 2012;8:8362. http://doi.org/10.15766/mep_2374-8265.8362
- [Background] Williams D, Fisicaro T, Hargraves R, Berg D. End-of-life communication education program for internal medicine residents. MedEdPORTAL Publications. 2009;5:7945. http://doi.org/10.15766/mep_2374-8265.7945
- [Result] Anspacher M, Shah N. Palliative care for the medically complex child. MedEdPORTAL Publications. 2013;9:9538. http://doi.org/10.15766/mep_2374-8265.9538